CLINICAL TRIAL: NCT05391113
Title: Stimuli Sociaux Et Non-sociaux Du Système De Récompense : Une Étude En IRM Chez Des Sujets Avec Trouble Du Spectre De L'autisme Et Des Sujets Avec Un Trouble Addictif À L'alimentation. - RESYSTAA
Brief Title: REward SYSTem in Autism Spectrum Disorder and Addictive Disorder
Acronym: RESYSTAA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Tours (Other)
Collaborators: INSERM UMR-1253, Tours, France (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: DR220016; 2022-A01098-35 (Registry Identifier: ID RCB-ANSM); 22-87 (Registry Identifier: CPP SUD-MED IV)
Record Dates: First submitted 2022-05-20; First posted 2022-05-25 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Autism Spectrum Disorder
Keywords: Autism; MRI;Addictive disorders
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder | interventions — Electroencephalography

STUDY DESIGN:
Intervention Model Description: Pilot study, monocentric open in three parallel groups (ASD, AD and healthy volunteers).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Autism Spectrum Disorder (Experimental): Characterized by two main diagnostic criteria: a socio-emotional deficit via a defect in communication and social reciprocity, and a behavioral deficit which manifests itself in repetitive behavioral patterns (stereotypes), restricted interests and/or activities.
  Interventions: Diagnostic Test: MRI; Diagnostic Test: EEG
- Food Addictive Disorders (Active Comparator): Characterized by regroup substance use disorders and behavioral addictions, are characterized in particular by the repeated occurrence of compulsive behavior and impaired social functioning
  Interventions: Diagnostic Test: MRI; Diagnostic Test: EEG
- Healthy volonteers (Placebo Comparator): Adult without neurological and psychiatric history, absence of progressive somatic pathologies or with vital risk.
  Interventions: Diagnostic Test: MRI; Diagnostic Test: EEG

INTERVENTIONS:
Diagnostic Test: MRI — an fMRI measurement of the BOLD physiological signal for sensory responses
  Other Names: Functionnal MRI
Diagnostic Test: EEG — These tests, through videos with a social or non-social content (human presence or absence on the stereoscopic projection), will allow us to study two types of sensorialities (visual and interoceptive). Thus, it will be possible to obtain inter- and exteroceptive profiles of the participants, a direct reflection of the processing of the internal bodily sensations of the body.
  Other Names: Electro Encephalography

SUMMARY:
An MRI Study in Subjects with Autism Spectrum Disorder and Subjects with Food Addictive Disorder compared to healthy volunteers.

DETAILED DESCRIPTION:
An MRI Study in Subjects with Autism Spectrum Disorder and Subjects with Food Addictive Disorder compared to healthy volunteers, where pathophysiology common to both disorders, based on a dysfunction of the reward system. The project we propose aims to explore the neural networks underlying these alterations in patients suffering from autism or addictive disorder.

ELIGIBILITY:
Inclusion Criteria:

Arm A ˗ Concerning ASD patients: Adult carrying the diagnosis of ASD (DSM-5, ADOS, ADI-R criteria)

Arm B ˗ Concerning FAD patients: Adult diagnosed with FA presenting with food addiction (DSM-5, YFAS 2.0, BES >= 18 criteria).

Arm C ˗ Concerning healthy volunteers : Adult with no neurological and psychiatric history , absence of progressive somatic pathologies or with vital risk.

For all participants:

* Age greater than or equal to 18 years old
* Without intellectual delay (IQ > 70).
* Able to understand and apply the instruction when an active task is proposed, according to the estimate of the investigator.
* Free, express, informed and written consent of the participant.
* Participant affiliated to a social security scheme

Exclusion Criteria:

* Neuromotor disorders.
* Visual disturbances not corrected or incompatible with MRI.
* Known epilepsy.
* Current substance use disorder with emotional distress/significant impact on functional outcome
* Rare genetic syndrome.
* Contraindications to MRI (other than body circumference)
* For women of childbearing age: negative urine or blood pregnancy test
* Person subject to a measure of judicial protection (safeguard of justice, curatorship, guardianship or family authorization)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2023-07-27 (Actual); Primary Completion 2026-07-27 (Estimated); Study Completion 2027-01-27 (Estimated)

PRIMARY OUTCOMES:
Blood Oxygene Level Dependent (BOLD) MRI signal | At inclusion
  Measurement in fMRI of the BOLD signal for each condition (interest, addiction, social) will be carried out in order to highlight the possible alterations of the reward system, in particular at the level of the striatum in terms of cerebral activation for each of the groups of subjects. (FAD, ASD and HV).

SECONDARY OUTCOMES:
Tolerance to an MRI examination for FAD with overweight or obesity | At inclusion
  For the tolerance to an MRI examination for FAD with overweight or obesity: feedback on their experience in MRI.
Regulation of sensory, an fMRI measurement of the BOLD physiological signal for sensory responses (sensory block) in terms of brain activation in patients | At inclusion
  Regulation of sensory, an fMRI measurement of the BOLD physiological signal for sensory responses (sensory block) in terms of brain activation in patients with FAD compared to ASD subjects and healthy volunteers.

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric BRIEND, PhD, Principal Investigator — University Hospital,Tours -INSERM U1253 iBrain
Locations (3):
- France (3):
  - Center-Val de Loire Region Autism Resource Center, Tours
  - University Addictology Service, Liaison Team and Addictology Care, Tours
  - University Hospital, Medical Imaging Service, Tours

IPD SHARING:
Plan to Share IPD: No